CLINICAL TRIAL: NCT03171285
Title: Risk of Cardiovascular Disease in Soccer Referees: a Cross Sectional Study
Brief Title: Cardiovascular Disease in Soccer Referees
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Other Study IDs: 038/2011
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Less than 35 years old: Clinical and laboratory evaluations
  Interventions: Other: Less than 35 years old
- Greater than or equal to 35 years: Clinical and laboratory evaluations
  Interventions: Other: Greater than or equal to 35 years

INTERVENTIONS:
Other: Less than 35 years old — Clinical and laboratory evaluations
  Groups: Less than 35 years old
Other: Greater than or equal to 35 years — Clinical and laboratory evaluations
  Groups: Greater than or equal to 35 years

SUMMARY:
Although the mortality rate among soccer players is low, it causes much impact on the entire community and is a fascinating conundrum. The aim of this study was to evaluate the cardiovascular risk of soccer referees, to describe the frequency of cardiovascular risk considering age groups younger and older than 35 years old and to relate the Framingham and PROCAM indices for the comparison of cardiovascular risk in soccer referees. 50 referees of Paulista Soccer Federation were subjected to clinical and laboratory based evaluations at the Center for Sports Health at the Faculty of Medicine of ABC, and divided into two groups: lower and higher than 35 years of age.

DETAILED DESCRIPTION:
This is a cross-sectional study performed in a non-probabilistic sample for convenience, derived from information collected from medical records of the Medical Statistics Service. Data were obtained through clinical evaluation information and subsidiary examinations of 50 high performance field soccer referees of the Paulista Soccer Federation (PFF), during a pre-season training period of the 2009 Brazilian soccer championship.

Emphasis was especially placed on exposure to risk factors for coronary artery disease, conceivably more responsible for sudden death, when congenital heart disease was excluded.

All subjects were acquiesced to clinical and laboratory evaluations at the Center for Health in Sport of the Faculty of Medicine of ABC (FMABC). The referees were split into two age groups, according to the median of their ages. One of the groups consisted of trained individuals < 35 years old while the other group was made up of referees > 35 years old.

Family history: Occurrence of one or more relatives with disease or death from cardiac disease aged less than 50 years; Report of cardiomyopathy, coronary artery disease, Marfan syndrome or long QT syndrome, severe cardiac arrhythmias, or other cardiovascular diseases.

Personal history: Syncope or pre-Syncope; Chest pain or discomfort; Lack of air or fatigue disproportionate to the effort made; Palpitations or irregular heartbeat.

Physical examination: Physical and/or ocular signs of Marfan Syndrome; Decreased femoral artery pulses or "tardus"; meso- or telo- systolic murmurs; Second abnormal heart sound (single or with fixed unfolding with breathing); Heart murmurs (grade 2/6 systolic or diastolic of any intensity); Irregular heart rate; Bilateral blood pressure greater than 140/90 mmHg in more than one measurement.

Biochemical tests: High density lipoprotein (HDL), low density lipoprotein (LDL), very low density lipoproteins (VLDL), triglycerides (TG) and fasting blood glucose levels (Glic) were analyzed. The biochemical blood tests were processed by the Clinical Laboratory of FMABC, certified by controlab and ANVISA. The reference standards were considered according to the Guidelines of the Brazilian Society of Cardiology.

Ergospirometry: The following parameters were analyzed: Ergospirometry (Ergo), Maximum heart rate (HRmax), Maximum oxygen consumption (VO2max) and Anaerobic threshold (LA). The ergospirometric data were obtained through the Centurion 200 Treadmill and Micromed® BRA ECG. Protocol: start with 10 km/h - 1% inclination and increase of 1 km every minute. Gas analyzer: Vmax, Encore 29 c, Sensormedics®, USA. Program 20-21. Gases in two torpedoes: (1) - oxygen (O2); 26% and (2) - Carbon Dioxide (CO2): 4%, oxygen (O2) = 16% and Nitrogen (N2).

Echocardiogram: Two-dimensional echocardiogram (ECO) with Doppler was obtained by Esaote® model AV3 Partner with 2.5 MHz transducer with color flow mapping.

Electrocardiogram: The electrocardiographic tracings were performed by the Ecafix® CardioPerfect 5.0 device coupled to a microcomputer with compatible HD and a 1.4 MB drive 60 Hz filter. Approved by the Food and Drug Administration (FDA), the records were taken at rest, on days when they had not performed exercises, and according to the best clinical practice. The interpretation of the ECG abnormalities was completed by an experienced specialist and according to the criteria established by Corrado et al., for which they were classified into two categories:

* Group 1: commonly observed in trained athletes (over 80%) sinus bradycardia, first-degree AV block, V1 notch QRS or incomplete right bundle branch block, early repolarization, LVH criteria according to voltage increase in V5 and V6 consistent with the athlete's age, ethnicity and degree of physical fitness, and which does not require additional testing.
* Group 2: less common ECG changes (less than 5%) and need to be better evaluated to exclude cardiovascular diseases: T-wave inversion, ST-segment depression, pathological Q-waves, left atrial enlargement, QRS shift to the left, left/right anterolateral hemiblock, right QRS deviation/left posterolateral lower hemiblock, right ventricular hypertrophy, complete left or right bundle branch block, long or short QT interval, early ventricular repolarization Brugada like, ventricular arrhythmias.

Framingham and PROCAM indexes The risk of developing cardiovascular disease is contingent on multiple variables that interrelate with each other, increasing the probability of developing atherosclerotic coronary disease. Each of the risk factors is assigned a value that reflects greater or lesser potential impact on the development of cardiovascular disease and the implementation of preventive measures, and likelihoods, when applied early, to avert the onset of this disease.

The Framingham risk index was constructed based on the Framingham study, a prospective observational survey developed in the small northeastern city of the United States of America. This study evaluated blood pressure, smoking, lipid profile and other characteristics of 5,300 individuals of different ethnicities residing in Framingham, aged between 30 and 74 years at the time of the initial observation, as well as their causes of death and disease.

This index analyzes the cardiovascular risk in relation to the chance of developing stroke, acute myocardial infarction and cardiovascular death for the subsequent 10 years. The Framingham cardiovascular risk index has the characteristic of categorizing the variables into a smaller number of sections or sections without significant differentiation of body mass, age, gender, total cholesterol, HDL, presence or absence of smoking and Diabetes Mellitus, systolic and diastolic blood pressure values. Total points represent the percentage of cardiovascular risk (acute myocardial infarction, stroke and cardiovascular death) in the following 10 years.

The PROCAM index is a cardiovascular risk index based on a European study that commenced in 1979 and was completed in 1985. A total of 5159 individuals, all males, aged 35 to 65 years. The PROCAM index identified the following variables: age, LDL-cholesterol, HDL-cholesterol, Triglycerides (this is the only criterion that considers it directly), smoking, Diabetes Mellitus, systolic blood pressure and family history (this variable is considered only by this risk score). The total points represent the risk of cardiovascular disease (acute myocardial infarction, stroke and cardiovascular death) in the ensuing 10 years.

ELIGIBILITY:
Inclusion Criteria:

* elite referees of the gold series of the Paulista Soccer Federation;
* registered for participation in the São Paulo professional soccer championship in 2009;
* eligible for pre-participative evaluation and have completed the entire series of tests considered indispensable for the present study.

Exclusion Criteria:

-

Ages: 25 Years to 44 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: 50 high performance field soccer referees of the Paulista Soccer Federation (PFF), during a pre-season training period of the 2009 Brazilian soccer championship.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-05-02 (Actual); Primary Completion 2009-12-12 (Actual); Study Completion 2009-12-12 (Actual)

PRIMARY OUTCOMES:
Higher risk for coronary artery disease in referees aged over 35 years old. | 7 months
  Higher risk for coronary artery disease in referees aged over 35 years old assessed by clinical and laboratory evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Artes,Ciencias e Humanidades da Universidade d Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided